CLINICAL TRIAL: NCT07294885
Title: Deep Cervical LymphatIc-Venous Anastomosis for Alzheimer's Disease (CLIVA-AD): a Prospective, Single-center, Randomized, Double Blinded Trial
Brief Title: Deep Cervical LymphatIc-Venous Anastomosis for Alzheimer's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Director, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Y (2025) 250
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LVA group (Experimental): patients will receive lymphaticovenous anastomosis
  Interventions: Procedure: deep cervical lymphaticovenous anastomosis
- Sham group (Sham Comparator): patients will undergo the LVA surgical procedure without performing the lymphaticovenous anastomosis.
  Interventions: Procedure: deep cervical lymphaticovenous anastomosis

INTERVENTIONS:
Procedure: deep cervical lymphaticovenous anastomosis — patients will receive deep cervical lymphaticovenous anastomosis

SUMMARY:
Lymphaticovenous anastomosis (LVA) is a microsurgical technique that involves anastomosing fine lymphatic vessels with adjacent veins to reestablish lymphatic drainage pathways. It is used in the treatment of lymphedema-related conditions and is characterized by minimal invasiveness and rapid recovery. Based on findings from animal studies, some physicians in China have attempted deep cervical lymphatic-venous anastomosis to improve intracranial lymphatic drainage in patients with Alzheimer's disease (AD). Most studies, including those from our center, have observed early postoperative improvements in various domains such as mood, memory, executive function, and communication abilities in the majority of patients. However, these symptomatic improvements are not sustained. The reasons for the early improvements remain unclear. Are they due to enhanced lymphatic drainage resulting from the surgery itself, or are they attributable to other factors such as anesthetic effects, vascular release, or modulation of sympathetic nerves? Therefore, it is necessary to conduct a randomized controlled trial with a sham surgery group to clarify the causes of early clinical symptom improvements. Based on this, this project aims to carry out a prospective, single-center, randomized double-blind controlled study to evaluate whether the early symptomatic improvements following deep cervical LVA in AD patients are attributable to the surgical intervention itself or to other aspects of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-80 years (inclusive), regardless of gender.
* Meeting the diagnostic criteria for Mild Cognitive Impairment or mild to moderate dementia due to Alzheimer's disease (according to the 2024 AA clinical diagnostic criteria for AD-related dementia).
* Disease duration of 6 months or longer, with no clinical improvement after 3 months or more of conservative treatment.
* MMSE score: 12-26.
* Biomarker confirmation of AD: positive Aβ-PET and tau-PET, or positive cerebrospinal fluid biomarkers.
* Having a reliable caregiver (providing companionship for ≥3 hours per day).
* Signed written informed consent from the patient or legally authorized representative.

Exclusion Criteria:

* Contraindications to MRI, ICG angiography, or PET.
* Contraindications to surgery or anesthesia, such as coagulation disorders (platelet count <100×10⁹/L, INR >1.7).
* Comorbid major organ dysfunction, such as reduced left ventricular ejection fraction, severe hepatic or renal insufficiency (AST or ALT >3 times the upper limit of normal; eGFR <30 mL/min/1.73m²).
* Intracranial structural lesions indicated by MRI, including brain tumors, cerebral infarction, intracranial hemorrhage, aneurysms, arteriovenous malformations, hydrocephalus, etc.
* MRI findings suggestive of significant cerebral small vessel disease features: more than one lacunar infarction in the deep white matter and periventricular regions and/or white matter hyperintensity (WMH) with a Fazekas grade >2, or the presence of ≥4 cerebral microbleeds.
* Other causes of dementia, such as hypothyroidism or vitamin B12 deficiency.
* Drug/alcohol addiction.
* Severe psychiatric illness or suicide risk.
* Comorbid medical conditions with a life expectancy of less than 1 year.
* Participation in another interventional trial within the past 3 months.
* Poor compliance or judged by the investigator as unsuitable for participation.
* Patients receiving therapy with Lecanemab or Donanemab.
* Other conditions that the researcher deems unsuitable for participation in this study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Montreal Cognitive Assessment (MoCA) score | 4±1 days
  MoCA ranges from 0 to 30, with higher score meaning better outcome
Changes in Mini-mental State Examination (MMSE) score | 4±1 days
  MMSE ranges from 0 to 30, with higher score meaning better outcome
Changes in Barthel index (BI) | 4±1 days
  BI ranges from 0 to 100, with higher score meaning better outcome
Changes in Clinician's Interview-Based Impression of Change-plus caregiver input (CIBIC-plus) | 4±1 days
  CIBIC-plus ranges from 1 to 7, with higher score meaning worse outcome

SECONDARY OUTCOMES:
Changes in Montreal Cognitive Assessment (MoCA) score | 90±7 days; 180±15 days; 270±20 days
  MoCA ranges from 0 to 30, with higher score meaning better outcome
Changes in Mini-mental State Examination (MMSE) score | 90±7 days; 180±15 days; 270±20 days
  MMSE ranges from 0 to 30, with higher score meaning better outcome
Changes in Barthel index (BI) | 90±7 days; 180±15 days; 270±20 days
  BI ranges from 0 to 100, with higher score meaning better outcome
Changes in Clinician's Interview-Based Impression of Change-plus caregiver input (CIBIC-plus) | 90±7 days; 180±15 days; 270±20 days
  CIBIC-plus ranges from 1 to 7, with higher score meaning worse outcome
Severe adverse events | Perioperative period